CLINICAL TRIAL: NCT01397591
Title: Phase II Trial of Ofatumumab and Bortezomib in Subjects With Relapsed Cluster of Differentiation Antigen 20 (CD20)+ Diffuse Large B Cell Lymphoma, Follicular Lymphoma, or Mantle Cell Lymphoma
Brief Title: Ofatumumab and Bortezomib in Subjects With Relapsed CD20+Diffuse Large B Cell, Follicular, or Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed by PI due to lower than expected accrual.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Millennium Pharmaceuticals, Inc. (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007042; NCI-2011-01032 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OFT113735 (Other: GlaxoSmithKline)
Record Dates: First submitted 2011-07-13; First posted 2011-07-19 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — ofatumumab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ofatumumab with Bortezomib (Experimental): Ofatumumab was given intravenously on cycle 1 day 1 at a dose of 300mg, followed by a cycle 1 day 8 dose of 1000mg. During cycles 2 through cycle 6, Ofatumumab was given at a dose of 1000mg on day 1 of each cycle, with no dosing on any other day of the cycle. Bortezomib was given intravenously at a dose of 1.6mg/m2 on days 1, 8, and 15 of each cycle, following the Ofatumumab infusion, if given.
  Interventions: Biological: Ofatumumab; Drug: Bortezomib

INTERVENTIONS:
Biological: Ofatumumab — Given intravenously
  Other Names: Arzerra; HuMax-CD20
Drug: Bortezomib — Given intravenously
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
This phase II trial studies how well giving ofatumumab together with bortezomib works in treating patients with relapsed diffuse large B cell lymphoma (DLBCL), follicular lymphoma (FL), or mantle cell lymphoma (MCL). Monoclonal antibodies, such as ofatumumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving ofatumumab together with bortezomib may help kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy, as measured by overall response (complete response (CR) + partial response (PR)) of ofatumumab in combination with bortezomib in subjects with relapsed cluster of differentiation (CD)20+ DLBCL, FL or MCL.

SECONDARY OBJECTIVES:

I. To explore duration of efficacy of ofatumumab in combination with bortezomib in the same population as measured by progression free survival (PFS), overall survival (OS) and disease free survival (DFS).

II. To assess response as compared to prior treatment. III. To assess the safety and tolerability of ofatumumab in combination with bortezomib in the same patient population.

TERTIARY OBJECTIVES:

I. Correlation of trough ofatumumab blood levels to response. II. Correlation fragment crystallizable receptor (FcR) gamma 3 allotype and response.

OUTLINE:

Patients receive ofatumumab intravenously (IV) over 2.5 hours on days 1 and 8 of course 1, and day 1 of all subsequent courses. Patients also receive bortezomib IV over 3-5 seconds on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy sample obtained within 6 months of study entry that:
* Is histologically confirmed DLBCL, MCL or FL, by an Oregon Health and Science University (OHSU) hematopathologist
* Retains expression of CD20+
* Patients must be refractory to or have recurrent disease after prior rituximab containing treatment; relapse or progression is defined according the International Working Group (IWG) response criteria
* FL patients must have disease-related symptoms, cytopenias, threatened end-organ function, bulky or progressive disease, or it is the patient's preference to be treated
* DLBCL and MCL patients must be either transplant ineligible or have refused high dose therapy
* Patients must have radiographically measurable disease, as defined by the IWG criteria; the same method of assessment used to measure each lesion at baseline must be used for all subsequent tumor measurements throughout the study
* There is no limit to the number of prior treatments
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 1.0 K/mm^3
* Platelets >= 50 K /mm^3
* Total bilirubin =< 1.5 x normal institutional limits, unless secondary to Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT))/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase (SGPT)) =< 2.5 x institutional upper limit of normal (ULN)
* Alkaline Phosphatase < 2.5 times ULN (unless due to disease involvement of the liver or bone marrow)
* Patients must be able to comply with study procedures and follow-up examinations
* Women of childbearing potential (not surgically sterile or < 12 months naturally post-menopausal) must be willing to use medically accepted method of contraception for the duration and 6 months following the end of the treatment; acceptable methods of contraception include abstinence, barrier method with spermicidal or hormonal contraceptive (oral, transdermal, implanted and injected) in conjunction with a barrier method
* Men who are not surgically sterile must practice abstinence or use a barrier method of birth control for the duration and 6 months following the end of treatment
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects who have current active hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Patients who have had chemotherapy, antibody or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C); corticosteroids for symptom control are allowed up to 7 days of starting protocol treatment
* Patients may not have received any other investigational agents within 4 weeks, or may not be currently participating in any other interventional clinical study
* Prior treatment with ofatumumab or bortezomib
* Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to start of therapy
* Diagnosis of another malignancy, unless the patient has been disease-free or at least 5 years following the completion of curative intent therapy with the following exceptions: patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed; patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ofatumumab or bortezomib
* Peripheral neuropathy or neuropathic pain of Grade 2 or greater
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or anti-viral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis and tuberculosis
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (New York Heart Association (NYHA) III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient
* Pregnant or breast feeding women
* Known human immunodeficiency virus (HIV) infection
* Positive serology for Hepatitis B (HB) defined as a positive test for HB surface antigen (HBsAg); in addition, if negative for HBsAG but HB core antibody (HBcAb) positive (regardless of HBsAb status), a HB deoxyribonucleic acid (DNA) test will be performed; if positive the subject will be excluded
* Active hepatitis C infection (HC) defined as a positive test for hepatitis C antibody (HCAb), in which case the investigator should reflexively perform a HC Recombinant Immunoblot assay (RIBA) on the same sample to confirm the result
* Known lymphoma involvement of the central nervous system (CNS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Okada, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects enrolled on study but 1 of the 3 was a screen failure so only 2 subjects were assigned to study treatment.
Groups:
- Ofatumumab in Combination With Bortezomib: All patients were given Ofatumumab in combination with Bortezomib in treatment cycles lasting 28 days. Ofatumumab was given intravenously on cycle 1 day 1 at a dose of 300mg, followed by a cycle 1 day 8 dose of 1000mg. During cycles 2 through cycle 6, Ofatumumab was given at a dose of 1000mg on day 1 of each cycle, with no dosing on any other day of the cycle. Bortezomib was given intravenously at a dose of 1.6mg/m2 on days 1, 8, and 15 of each cycle, following the Ofatumumab infusion, if given.
Period: Overall Study
Arm/Group | Ofatumumab in Combination With Bortezomib
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab in Combination With Bortezomib
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Ofatumumab in Combination With Bortezomib in Patients With Relapsed CD20+ (Cluster of DIfferentiation Antigen 20) Diffuse Large B Cell Lymphoma, Follicular Lymphoma, or Mantle Cell Lymphoma
Description: Based on International Working Group (IWG) criteria, recorded in four categories: Complete Response (CR), disappearance of all evidence of disease; Partial Response (PR), regression of measurable disease and no new sites of disease; Progressive Disease (PD), Any new lesion or increase by >= 50% of previously involved sites from nadir. Stable Disease (SD), failure to attain CR/PR or PD. A response is defined to be either CR/PR. A failure in response includes SD/PD.
Time Frame: Every 2 cycles during treatment and then every 3 months for 2 years
Measure: Number; unit: participants
Groups:
- Treatment (Monoclonal Antibody and Enzyme Inhibitor Therapy): Patients receive ofatumumab IV over 2.5 hours on days 1 and 8 of course 1, and day 1 of all subsequent courses. Patients also receive bortezomib IV over 3-5 seconds on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  ofatumumab: Given IV
  bortezomib: Given IV
  laboratory biomarker analysis: Correlative studies
  enzyme-linked immunosorbent assay: Correlative studies
  biopsy: Optional correlative studies
  quality-of-life assessment: Ancillary studies
  polymorphism analysis: Correlative studies
  flow cytometry: Correlative studies
Arm/Group | Treatment (Monoclonal Antibody and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: Overall Survival
Description: This outcome measure is defined as the time from initiation of treatment to death due to any cause.
Time Frame: Up to every 3 months for 2 years
Population: Study closed by PI due to lack of accrual before this outcome measure could be analyzed.
Arm/Group | Treatment (Monoclonal Antibody and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival
Description: This outcome measure is defined as the length of time after treatment during which the patient survives with no sign of the disease.
Time Frame: Up to every 3 months for 2 years
Population: Study closed by PI due to lack of accrual before this outcome measure could be analyzed.
Arm/Group | Treatment (Monoclonal Antibody and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Disease Free Survival
Description: The period of time between complete remission and recurrence of disease.
Time Frame: Up to every 3 months for 2 years
Population: Study closed by PI due to lack of accrual before this outcome measure could be analyzed.
Groups:
- Ofatumumab in Combination With Bortezomib: All patients were given Ofatumumab in combination with Bortezomib in treatment cycles lasting 28 days. Ofatumumab was given intravenously on cycle 1 day 1 at a dose of 300mg, followed by a cycle 1 day 8 dose of 1000mg. During cycles 2 through cycle 6, Ofatumumab was given at a dose of 1000mg on day 1 of each cycle, with no dosing on any other day of the cycle. Bortezomib was given intravenously at a dose of 1.6mg/m2 on days 1, 8, and 15 of each cycle, following the Ofatumumab infusion, if given.
  ofatumumab: Given IV
  bortezomib: Given IV
  laboratory biomarker analysis: Correlative studies
  enzyme-linked immunosorbent assay: Correlative studies
  biopsy: Optional correlative studies
  quality-of-life assessment: Ancillary studies
  polymorphism analysis: Correlative studies
  flow cytometry: Correlative studies
Arm/Group | Ofatumumab in Combination With Bortezomib
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Adverse Events (Toxicity)
Description: Toxicities and adverse experiences will be assessed at each visit using the NCI Common Toxicity Criteria for Adverse Events v4.0 Interim analyses on toxicity will be implemented based on the toxicity endpoints of the first 6 patients, and will be conducted sequentially 4 weeks after the treatment of each patient, or when serious toxicity has been observed for the patient, whichever comes earlier. we assume a non-informative prior distribution (Beta (0.001, 0.001)) for toxicity rate, and compute the posterior distribution of toxicity rate sequentially.
Time Frame: Days 1, 8, and 15 of each course and 4-6 weeks after final treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Monoclonal Antibody and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Arm/Group | Ofatumumab in Combination With Bortezomib
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab in Combination With Bortezomib (N=2)
Nausea (Gastrointestinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Infusion Reaction (Immune system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Sensory Neuropathy (Nervous system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Upper GI Hemorrhage (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Laryngeal Inflammation (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Memory Impairment (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No